CLINICAL TRIAL: NCT02094404
Title: Triage of Children at the Emergency Department: Manchester Triage System or Pediatric Early Warning Score?
Status: Completed | Type: Observational
Sponsor: E.P. de Groot (Other)
Responsible Party: Sponsor-Investigator, E.P. de Groot, MD, Isala
Organization: Isala (Other)
Other Study IDs: KSEH13
Record Dates: First submitted 2014-03-08; First posted 2014-03-21 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Triage of Children
Keywords: Emergency Department; Pediatric Early Warning Score; Manchester Triage System
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children at the ED<18yr

SUMMARY:
Currently, the Manchester Triage System (MTS) is used to triage all children presenting at the emergency department(ED) in this hospital. This system has been proven safe, but many patients are classified as too urgent. In this hospital adults are prioritised at the ED by a score based on vital signs, the early warning score. A similar score is developed suitable for children. This score, the Pediatric Early Warning Score (PEWS), is already used to determine clinical deterioration.

The investigators hypothesize that children can be triaged safely with the PEWS.

If it is safe, there will be one triage system again at the ED. Another advantage will be more continuity in assessing the condition of patients who are admitted to the hospital.

DETAILED DESCRIPTION:
Background: Triage systems are used at EDs to prioritize patients to make sure that those who need it, receive immediate care.

The MTS is used for children at EDs by many hospitals worldwide, also at the ED of the Isala, the Netherlands. This triage system has been proven safe, but many patients are classified as too urgent. This is a disadvantage because accurate triage is needed to provide access for immediate ill patients and for sufficient flow at the ED.

Currently, adult patients at the ED of the Isala are classified by the early warning score. This is a score based on vital signs and it is easily calculated. It originally has been developed to determine clinical deterioration. For children normal values are different for each age. Therefore there has been developed the PEWS, which is now only used to evaluate clinical patients. Ideally for the continuity in this hospital, there would be one system which can be used for triage as well as for clinical patients. The investigators hypothesize that the PEWS is a safe alternative for the triage of children at the ED.

Design: A form will be attached on the file of all children presenting at the ED, for recording data. These forms will be collected afterwards. The emergency department nurses will record the vital signs, which the investigators need to calculate the PEWS as well as the urgency determined by the MTS for each patient. The expert opinion will also be recorded. This is de urgency according to the doctor who has seen the patient, maximal acceptable door-to-doctor time: very urgent (immediate), urgent (<15minutes) or normal (<1hour). At the end of the consultation at the ED, the reference standard will be determined for each patient independent of MTS urgency or PEWS, with data available from the patient file. (1) For secondary outcome measures may or may not hospital admission or intensive care admission will be recorded.

No interventions are made and this study is of no influence on the treatment of the patients.

ELIGIBILITY:
Inclusion Criteria:

* All children presenting at the Emergency Department of the Isala.

Exclusion Criteria:

* Children seen in room 17, the plaster and little trauma room (because of practical reasons).

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: - All children presenting at the emergency department of the Isala, Zwolle.
Sampling Method: Non-Probability Sample
Enrollment: 727 (Actual)
Dates: Start 2013-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Reference standard | <1day
  A reference standard as developed by van Veen et al with 5 urgency levels to be determined with the information available from the patient file as documented after presentation at the ED.
  The reference standard will be separately compared to the MTS as well as the PEWS as determined for each patient presenting at the ED.

SECONDARY OUTCOMES:
Hospital admission | <12 hours
  Hospital or intensive care admission directly following visiting the ED or to the utmost <12h.
  Admission: yes/no.

OTHER OUTCOMES:
Expert opinion | <10 minutes
  Assessed directly at the first contact with the patient at the ED by the pediatrician. Maximal acceptable door-to-doctor time: very urgent (immediate), urgent (<15minutes) or normal (<1hour).

CONTACTS AND LOCATIONS:
Overall Officials: E.P de Groot, MD, Principal Investigator — Isala
Locations (1):
- Isala, Zwolle, Overijssel, Netherlands

REFERENCES:
- [Background] van Veen M, Steyerberg EW, Ruige M, van Meurs AH, Roukema J, van der Lei J, Moll HA. Manchester triage system in paediatric emergency care: prospective observational study. BMJ. 2008 Sep 22;337:a1501. doi: 10.1136/bmj.a1501. PMID 18809587